CLINICAL TRIAL: NCT01042275
Title: Patient-reported Mid- and Long-term Outcome After Insertion of Retropubic and Transobturator Tapes Using the Incontinence Outcome Questionnaire (IOQ)
Brief Title: Patient-reported Outcome After Sling Insertion Using the Incontinence Outcome Questionnaire (IOQ)
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: FHKUZH10-2008
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2010-04

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; retropubic sling; transobturator sling; tension-free vaginal tape; transobturator tape; TVT; TVT-O; TOT; REMEEX; IVS
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- TOT: transobturator sling, outside-in (TOT)
- TVT-O: Tension-free transobturator tape, inside-out (TVT-O)
- IVS: retropubic Intravaginal Sling (IVS)
- TVT: retropubic tension-free vaginal tape (TVT)
- REMEEX: Re-adjustable mechanical external sling (REMEEX)

SUMMARY:
Midurethral tapes are by now standard procedure in the surgical treatment of women with stress urinary incontinence. While the retropubic TVT is well documented with long-term results up to 11 years and continence rates of 90 %, the published data for the transoburator tapes (TO) cover follow-up of 3 years only. So far, all tapes establish continence effectively. Recently, the detailed 27-item Incontinence Outcome Questionnaire (IOQ) was constructed to assess patient-reported outcome and quality of life after insertion of a midurethral tape and validated for the German language. The aim of this study was to evaluate patient-reported mid- and long-term outcome after insertion of tension-free vaginal tape (TVT), transobturator sling, outside-in (TOT) and tension-free transobturator tape, inside-out (TVT-O).

ELIGIBILITY:
Inclusion Criteria:

* incontinence sling
* time frame 1/1999 - 12/2007

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were treated at 2 Swiss public teaching hospitals
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
patient's satisfaction | 3/2009

SECONDARY OUTCOMES:
re-admission | 3/2009

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Betschart, MD, Principal Investigator — Clinic for Gynecology, University Hospital of Zurich
Locations (1):
- University of Hospital, Clinic for Gynecology, Zurich, Switzerland